CLINICAL TRIAL: NCT07274241
Title: Escitalopram Dose and the Risk of Serious Adverse Events in Older Adults With Low Kidney Function: A Population-Based Cohort Study Research Protocol
Brief Title: Escitalopram and the Risk of Serious Adverse Events
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 2025 0906 615 000; ICES # 2025 0906 615 000 (Other: ICES)
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease (CKD); Elderly; Outpatient
Keywords: Chronic Kidney Disease; High-throughput computing; Drug Adverse Events; Selective Serotonin Reuptake Inhibitors; Escitalopram; Elderly; Geriatrics; Drug Safety
MeSH Terms: conditions — Renal Insufficiency, Chronic; Drug-Related Side Effects and Adverse Reactions | interventions — Escitalopram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low dose of Escitalopram (5 mg/day): Residents of Ontario (and possibly Alberta), aged 66 years or older with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for Escitalopram (low-dose 5 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to January 1, 2025, with a day supply of ≥7 days. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, and each patient will enter the cohort only once.
  Interventions: Drug: Escitalopram
- High dose of Escitalopram (10 mg/day): Residents of Ontario (and possibly Alberta), aged 66 years or older with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new oral prescription for Escitalopram (high-dose: 10 mg/day) at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program from January 01, 2008, to January 1, 2025, with a day supply of ≥7 days. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, and each patient will enter the cohort only once.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — The primary exposure of interest will be oral Escitalopram at a dose of 5 or 10 mg/day.

SUMMARY:
The goal of this population-based cohort study is to assess the safety of initiating a new outpatient prescription of 10mg/day of Escitalopram (higher dose) compared to 5 mg/day (lower dose) in adults over the age of 65 with low kidney function.

Primary question

Whether initiating a new outpatient prescription of a higher dose of Escitalopram (10mg/day) compared to a lower dose (5 mg/day) in older adults with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) is associated with a higher 30-day risk of a composite outcome of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality?

DETAILED DESCRIPTION:
Background Many older adults experience mental health disorders, such as depression and anxiety, alongside having low kidney function. Escitalopram, a selective serotonin reuptake inhibitor, is a commonly prescribed antidepressant to older adults for depression and anxiety treatment, but aging and low kidney function can lead to increased plasma levels and a higher risk of adverse events. Inconsistent starting dose adjustments for patients with low kidney function have been noted in prescribing references, product monographs, and other standard sources. This may be one reason for the inconsistent dosing observed in routine practice, where many older adults with low kidney function are initiated on escitalopram at a dose of 10 mg per day. Such a dose, compared to the lower dose of 5 mg per day, may be associated with a higher rate of falls, fractures, gastrointestinal bleeding, arrhythmias, hospitalization, and mortality. Despite these concerns, there is a lack of real-world evaluation.

Using a novel high-throughput approach using Ontario healthcare databases, the investigators identified an increased risk of adverse outcomes in patients with advanced CKD (estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m² without a history of dialysis or a kidney transplant) who were newly prescribed Escitalopram compared to a similar cohort of non-users.

To advance and validate these early findings, the investigators plan to conduct a population-based retrospective cohort study among older adults in Ontario, Canada. This study will use data to investigate the 30-day risk of serious adverse events after starting high versus low doses of escitalopram in older adults with low kidney function, aiming to enhance safer prescribing practices.

Methods

In this population-based retrospective cohort study, eligible participants will include older adults (≥66 years) with eGFR <45 mL/min/1.73 m2 (not receiving dialysis or having a history of kidney transplantation) from Ontario (and possibly Alberta) who were dispensed a new outpatient prescription for oral Escitalopram (5 or 10 mg/day) with a day supply of ≥7 days. In Ontario, accrual will occur between January 1, 2008, and January 1, 2025. Based on the prescribed daily dose, individuals will be divided into two groups: low-dose (5 mg/day) and high-dose (10 mg/day). Propensity score weighting will be used to ensure both groups are well-balanced on a comprehensive set of measured baseline characteristics. The primary outcome will be a 30-day composite of all-cause hospitalization, emergency department visit, or mortality.

Objectives

Is there a higher 30-day risk of a composite outcome of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality among older adults with low kidney function (an eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who initiate a high dose (10 mg/day) versus a low dose (5 mg/day) escitalopram in the outpatient setting?

Does the category of baseline eGFR modify the risk of a 30-day composite outcome, , among patients who initiate a higher dose versus a lower dose of escitalopram in the outpatient setting? The cohort will be expanded to include all levels of baseline eGFR, and eGFR will be categorized as ≥60, 45-59, and <45 mL/min per 1.73 m².

Study Design and Setting

Data Sources: The investigators propose a population-based retrospective cohort study using using linked administrative health data from Ontario, Canada. If the Ontario cohort is small to generate reliable estimates, the investigators will augment the sample size by performing the same analysis using Alberta health administrative data.

Ontario data will be sourced from ICES (ices.on.ca). It offers secure, encrypted individual-level data for Ontario residents, all with universal access to hospital and physician services under a government-funded, single-payer healthcare system. The use of data in this study is authorized under section 45 of Ontario's Personal Health Information Protection Act, which does not require review by a research ethics board. The study will use Ontario's comprehensive health databases, such as the Ontario Drug Benefit (ODB) for prescription data, the Registered Persons Database (RPDB) for demographics and vital status, Canadian Institute for Health Information Discharge Abstract Database (CIHI-DAD)and National Ambulatory Care Reporting System (NACRS) for hospitalizations and emergency visits, Ontario Health Insurance Plan (OHIP) Database for physician billing claims, and Ontario Laboratories Information System (OLIS) for laboratory data, including serum creatinine, to estimate kidney function.

If the investigators proceed with conducting the study in Alberta, the Alberta data will be accessed through the Alberta Kidney Disease Network (AKDN). This dataset ends in ~ 2021.

The investigators are publicly registering the study protocol and documenting the study description, design, and statistical analysis prior to conducting outcome analyses. The results of this study will be reported adhering to RECORD reporting guidelines.

Study Population

The investigators will include all older adults (≥66 years) with an eGFR <45 mL/min per 1.73 m2 (not receiving dialysis or having a history of kidney transplantation) who received a new outpatient prescription for oral escitalopram with an initial dose of 5 or 10 mg/day and a day supply of ≥7 days between 2008 and 2024. The dispensing date of the prescription will serve as the index date, and only the first eligible prescription will be included to ensure unique cohort entry. Each individual can enter the cohort only once. Patients will be categorized into "high-dose" and "low-dose" SSRI users.

Baseline Characteristics

Health records, census files, hospital records, laboratory data, and physician claims will provide baseline variables, including demographic characteristics (such as age, sex, rurality, and neighborhood income quintile), comorbidities, and medication use. Baseline comorbidities and healthcare utilization will be assessed using 5-year and 1-year look-back periods from the index date, respectively. Baseline medication use will be assessed within 120 days prior to the index date. Patients are required to have an outpatient serum creatinine level measured within 365 days prior to cohort entry, allowing for the estimation of eGFR using the 2021 CKD-EPI equation. Exclusion criteria include end-stage kidney disease (on dialysis or having received a kidney transplant).

Outcomes

The prespecified primary outcome is defined as the 30-day composite outcome of all-cause hospitalization, emergency department visit, or mortality. Only the first hospitalization or emergency department visit in the first 30 days is counted. The components of the primary composite outcome (all-cause hospitalization, all-cause emergency department visits, or all-cause mortality) is accurately coded in ICES data. The observation window for study outcomes will begin on the date of prescription fill and will last 30 days post-initiation. Loss to follow-up for study outcomes is expected to be <0.3% as the observation window for outcomes will be <90 days, and provincial emigration in this age group (the only reason for loss to follow-up) is <0.5% annually. Participant observation time will be censored at the time of the first occurrence of the outcome of interest, death (if not the outcome of interest), or 30 days after the index date, whichever comes first.

Secondary outcomes will include

1. Components of the primary composite outcome: 30-day all-cause hospitalization, all-cause emergency department visit, and all-cause mortality, each of which is examined separately.
2. 30-day composite outcome of a hospital encounter (hospital admission or emergency department visit) with delirium or encephalopathy (disorientation, transient alteration of awareness, other and unspecified symptoms and signs involving cognitive function) or hospital encounter with receipt of an urgent computed tomography scan of the head.
3. 30-day composite outcome of a hospital encounter (hospital admission or emergency department visit) with fracture (hip, femur, humerus, wrist/forearm, pelvis, and spine), falls, hypotension, or syncope
4. 30-day hospital encounter (hospital admission or emergency department visit) with composite outcome of atrial fibrillation/flutter or ventricular arrhythmia, or other arrhythmia (including pacemaker insertion, palpitations, tachycardia unspecified, atrioventricular block, supraventricular tachycardia, other conduction disorders, implantable cardiac defibrillator)

Statistical analysis plan

Categorical variables will be summarized as frequencies and proportions, while continuous variables will be summarized as means with standard deviations (SD) or medians with interquartile ranges (IQR), as appropriate.

Baseline characteristics will be compared between the groups, starting with the high-dose (10 mg/day) and the low-dose (5 mg/day) groups, using standardized mean differences (SMDs). An absolute SMD greater than 10% will be considered indicative of a meaningful imbalance.

Balancing comparator group: The investigators will use inverse probability of treatment weighting (IPTW) on the propensity score to balance baseline characteristics between the high-dose (10 mg/day) and low-dose (5 mg/day) groups, including known predictors of escitalopram use. Propensity scores will be generated using a multivariable logistic regression model with all baseline characteristics. The average treatment effect in the treated (ATT) weights will be used, where patients in the low-dose group will be assigned weights calculated as (propensity score / [1 - propensity score]), and patients in the high-dose group will receive a weight of 1. This method will produce a weighted pseudo-sample of patients in the referent group, i.e., low-dose escitalopram (5 mg/day), with a similar distribution of measured baseline characteristics as the high-dose escitalopram (10 mg/day) group. Baseline characteristics will be compared between groups using standardized differences in both unweighted and weighted samples.

Regression analysis: To evaluate the primary outcome composite measure of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality, the investigators will apply a modified Poisson regression analysis to estimate the risk ratio (95% CI) and binomial regression to estimate the risk difference (95% CI) using the weighted cohort, with the low-dose escitalopram (5 mg/day) group as the referent.

Secondary analyses: The investigators will conduct independent testing for all secondary outcomes without adjusting for multiple comparisons. Each test will be performed and reported independently.

In line with best practices, the primary outcome will be presented with its P-value, and the investigators will report all secondary outcomes using point estimates with 95% confidence intervals.

Additional analyses

The investigators plan to conduct five additional analyses.

1. Effect measure modification (EMM): For EMM, the investigators will expand the cohort to all the eGFR levels and categorize them into three groups: eGFR ≥60, 45-<60, and <45 mL/min/1.73 m2. Baseline characteristics between high-dose (10 mg/day) and low-dose (5 mg/day) escitalopram groups will be assessed using standardized differences for all renal function categories combined and then within each of three eGFR categories (≥60, 45-<60, and <45 mL/min/1.73 m²).

   To balance baseline characteristics between high-dose and low-dose escitalopram groups, the investigators will apply the IPTW method (described above), based on propensity scores for all the eGFR categories combined and within each of the three eGFR categories.

   EMM will be assessed on both the additive and multiplicative scales.
   * For additive interaction, the investigators will use binomial regression with an identity link to estimate risk differences, including an interaction term between low-dose and high-dose escitalopram groups and eGFR strata.
   * For multiplicative interaction, the investigators will use modified Poisson regression analysis to estimate risk ratios, including an interaction term between low-dose and high-dose escitalopram groups and eGFR strata.
2. The high-throughput computing analysis in which the investigators executed 700+ population-based, new-user cohort studies, each comparing 74 acute (30-day) outcomes across strata of kidney function (PMID: 38186562) suggested escitalopram use versus no use causes harm in patients with low kidney function. The high-throughput computing analysis used Ontario data from January 1, 2008 to March 1, 2020. A subgroup analysis will be performed for the primary analysis restricting the cohort to before March 1, 2020 (overlap with high-throughput computing period) and after March 1, 2020 (no overlap).
3. Compute the hazard ratio for all outcomes within 30 days, illustrating the effect of the intervention on each outcome over time. The investigators expect hazard ratios to be similar to risk ratios.
4. Perform E-value analyses to determine the minimum association strength an unmeasured confounder would need with both the prescription drug and the outcome of interest to eliminate the observed association.
5. The investigators will compare risk of the primary outcome between a group of new users of 10 mg/day of escitalopram vs. a group of older adults with no escitalopram use (non-users). The same will also be done with a group of new users of 5 mg/day of escitalopram vs. a group of older adults with no escitalopram use (non-users). The investigators will utilize the same baseline characteristics, and employ the statistical analysis methods used in the primary analysis.

Combining Outcome Results from Ontario and Alberta

*This approach will only be used if the investigators proceed with analyzing Alberta data.

Privacy-preserving methods:

In Canada, the investigators are unable to connect individual-level patient data from different provinces due to privacy concerns. However, the investigators will combine results from both provinces (Ontario and Alberta) using a privacy-preserving method, to maintain data privacy and regulatory compliance. The proposed method requires only a single transfer of summary-level outputs from each province to the research team (will be adapted from the techniques of Shu et al. 2025).

ELIGIBILITY:
Inclusion Criteria:

* Older adult aged 66 years or greater with low kidney function (an eGFR <45 mL/min per 1.73 m2 ) who have filled a new oral prescription for Escitalopram at an outpatient pharmacy under the Ontario Drug Benefit (ODB) program with a dose of 5 or 10 mg/day and a day supply of ≥7 days from January 1, 2008, to January 1, 2025 for Ontario (if needed, dates in Alberta to be finalized based on data availability). The investigators will exclude individuals undergoing dialysis or those who have received a kidney transplant. The age criterion is set to guarantee that individuals in this population had at least one year of prior universal outpatient prescription drug coverage. The date when the prescription was filled will serve as the patient's entry or index date for the cohort, with each patient entering the cohort only once.

Exclusion Criteria:

1. Individuals with missing administrative database number, missing or invalid age (<0 or >105 years), missing or invalid sex, death on or before the index date, non-Ontario resident (for Ontario data).
2. Individuals less than 66 years of age on the index date.
3. Those with evidence of any study drug prescription 180 days before the index date (to restrict to new users only).
4. Individuals with other Selective Serotonin Reuptake Inhibitors (Citalopram, Fluoxetine, Fluvoxamine, Paroxetine, Sertraline) prescription in the previous 180 days before the index date or on the index date.
5. Individuals with more than one study drug prescription on the index date, as this complicates the ability to ascertain the prescribed dose accurately.
6. Individuals with end-stage renal disease, chronic dialysis, or a kidney transplant prior to the index date.
7. Evidence with hospital discharge or emergency department visit in the two days prior to or on the index date to ensure a new outpatient prescription.
8. Individuals with no serum creatinine lab value in the 0-365 days prior to the index date.
9. Individuals with unstable baseline kidney function:

   * If the most recent serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] (refer to this as test date 1), and there is not at least one 'outpatient' serum creatinine in the year before test date 1, OR
   * If the most recent prior serum creatinine test prior to the index date was an inpatient test [ER or hospitalization] (refer to this as test date 1), and while there is at least 'outpatient' serum creatinine test in the year before (test date 1), the most recent outpatient test prior to (test date 1) differs by an eGFR 10 mL/min/1.73 m2 or more from the value on (test date 1).

   In Ontario, it has been shown that an outpatient serum creatinine measurement in the province, conducted on a single occasion, usually represents a stable value.
10. Individuals receiving palliative care in the year prior to the index date, as in this setting dosing is less relevant; rather, the focus is comfort care.

The investigators will restrict to the first prescription in individuals with more than one eligible prescription. Date of this prescription will be the index date (the date from which the outcomes start being assessed).

Min Age: 66 Years | Sex: All
Age Groups: Older Adult
Study Population: Adults aged 66 years or older with low kidney function (eGFR <45 mL/min per 1.73 m2 but not receiving dialysis or having a history of kidney transplantation) who have filled a new outpatient prescription for Escitalopram with a dose of 5 or 10 mg/day and a day supply of ≥7 days between 2008 and 2024 in Ontario. The study accrual period for Alberta (if needed) will be determined based on data availability.
Sampling Method: Non-Probability Sample
Enrollment: 12145 (Actual)
Dates: Start 2008-01-01; Primary Completion 2025-01-01 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
A composite outcome of all-cause hospitalization, all-cause emergency department visit, or all-cause mortality. | Older adults exposed to high-dose (10mg/day) vs low-dose (5 mg/day) Escitalopram between Jan 1, 2008, and Jan 1,2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  All-cause hospitalization, all-cause emergency department visits, and all-cause mortality will be combined into a composite measure. Only the first hospitalization or first emergency department visit occurring after the cohort entry date will be considered.

SECONDARY OUTCOMES:
All-cause hospitalization | Exposed cohort to Escitalopram (high dose (10mg/d) versus low dose (5 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause hospitalization, individually presented as a secondary outcome. Only the first hospitalization after the cohort entry date will be considered.
All-cause emergency department visit | Exposed cohort to Escitalopram (high dose (10mg/d) versus low dose (5 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause emergency department visit, individually presented as a secondary outcome. Only the first emergency department visit after the cohort entry date will be considered.
All-cause mortality | Exposed cohort to Escitalopram (high dose (10mg/d) versus low dose (5 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  One of the components of the primary composite outcome, all-cause mortality, individually presented as a secondary outcome.

OTHER OUTCOMES:
30-day hospital encounter with composite outcome of Atrial Fibrillation/flutter or ventricular arrhythmia or other arrhythmia | Exposed cohort to Escitalopram (high dose (10mg/d) versus low dose (5 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  30-day hospital encounter (hospital admission or emergency visit) composite of atrial fibrillation/flutter or ventricular arrhythmia, or other arrhythmia (including pacemaker insertion, palpitations, tachycardia unspecified, atrioventricular block, supraventricular tachycardia, other conduction disorders, implantable cardiac defibrillator)
30-day composite outcome of a hospital encounter with delirium, encephalopathy, or hospital encounter with receipt of an urgent computed tomography scan of the head | Exposed cohort to Escitalopram (high dose (10mg/d) versus low dose (5 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with delirium or encephalopathy (disorientation, transient alteration of awareness, other and unspecified symptoms and signs involving cognitive function) or hospital admission with receipt of an urgent computed tomography scan of the head.
30-day composite outcome of a hospital encounter with fracture, falls, hypotension, or syncope | Exposed cohort to Escitalopram (high dose (10mg/d) versus low dose (5 mg/d)) between January 1, 2008, and January 1, 2025 will enter the cohort and will be followed until study outcome (first event), death, or 30 days from the cohort entry date.
  30-day composite outcome of a hospital encounter (hospital admission or emergency visit) with fracture, falls, hypotension, or syncope.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Garg, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute
Locations (1):
- London Health Sciences Centre Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The dataset in Ontario from this study is held securely in coded form at ICES. While legal data sharing agreements between ICES and data providers (e.g., healthcare organizations and government) prohibit ICES from making the dataset publicly available, access may be granted to those who meet pre-specified criteria for confidential access, available at www.ices.on.ca/DAS (email: das@ices.on.ca). The full dataset creation plan and underlying analytic code are available from the authors upon request, understanding that the computer programs may rely upon coding templates or macros that are unique to ICES and are therefore either inaccessible or may require modification.

REFERENCES:
- [Background] Abdullah SS, Rostamzadeh N, Muanda FT, McArthur E, Weir MA, Sontrop JM, Kim RB, Kamran S, Garg AX. High-Throughput Computing to Automate Population-Based Studies to Detect the 30-Day Risk of Adverse Outcomes After New Outpatient Medication Use in Older Adults with Chronic Kidney Disease: A Clinical Research Protocol. Can J Kidney Health Dis. 2024 Jan 6;11:20543581231221891. doi: 10.1177/20543581231221891. eCollection 2024. PMID 38186562